CLINICAL TRIAL: NCT03673917
Title: Cosmetology Students and Skin Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Principal Investigator, Lori Fischbach, Associate Professor of Epidemiology, University of Arkansas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 205582
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Intervention Model Description: The study design protocol is as follows: Schools of cosmetology in Arkansas are randomized using simple randomization to receive either 1) our educational video on skin cancer for cosmetologists or 2) a publicly accessible healthy lifestyle video on YouTube, which does not contain any information on skin cancer. Students view the video that was randomly assigned to the school they attended. Pre-video tests are administered at the school during classes or online at the students' convenience; the video intervention follows immediately, also during classes or online. Post-video test (in class or online) are administered 3 to 6 months after watching the video. All schools continued to also use their previous educational materials on skin cancer concurrent with our program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational video (Experimental): The educational video on skin cancer for cosmetologists
  Interventions: Other: Educational video
- Control video (Active Comparator): A publicly accessible healthy lifestyle video on YouTube, which did not contain any information on skin cancer
  Interventions: Other: Control video

INTERVENTIONS:
Other: Educational video — The educational video on skin cancer for cosmetologists
  Arms: Educational video
Other: Control video — A publicly accessible healthy lifestyle video on YouTube, which does not contain any information on skin cancer
  Arms: Control video

SUMMARY:
Assess the efficacy of training cosmetology students to detect suspicious skin lesions.

DETAILED DESCRIPTION:
The incidence of melanoma is increasing the USA. The early detection of skin cancer is associated with a significant decrease in morbidity and mortality. Hair professionals (cosmetologists and barbers) have an excellent opportunity to detect suspicious skin lesions on the scalp, neck, and face due to routinely looking at this area during customer visits. Currently in Arkansas, cosmetology schools teach students about how to recognize skin cancer on their clients. In this program, the aim was to improve the educational module for skin cancer in schools of cosmetology in Arkansas. In the proposed study, the intervention training module was designed to increase the knowledge of cosmetology schools students about skin cancer will be evaluated. It was hypothesized that this educational video will educate cosmetology students and cosmetologists about how to prevent skin cancer, how to recognize a suspicious spot or mole which may be a skin cancer, and how to talk with clients about seeing a dermatologist when a suspicious spot is found. This study was a cluster-randomized controlled trial in cosmetology schools in Arkansas. The institutional review board for human subjects at the University of Arkansas for Medical Sciences determined that this study was approved as exempt and submission was not required since it was an educational intervention to improve the quality of an educational component of the existing curriculum.

ELIGIBILITY:
Inclusion Criteria:

* For Schools: the school director agrees to participate and provide written consent
* For Students: Students were eligible at the enrolled schools if they agreed in writing to participate, filled out the baseline questionnaire, and viewed the assigned video.

Exclusion Criteria:

* The school had not recently or was not currently implementing a similar program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Students' knowledge | 3 - 6 months
  Scale name: Change in students' scores for knowledge of skin cancer, risk factors, and recognizing an abnormal skin spot. What scale measures: Scores were computed as the proportion of questions that the student correctly answered, and change in scores was computed by subtracting the pre-test score from the post-test score. If a student correctly answered a greater proportion of questions on the post-test compared to the pre-test, then they would have a positive value for the change in scores, and would be classified as increasing their knowledge. Scale ranges: The change in scores range from -100% to 100%; a change >0% is considered to be an increase in score and a better outcome, whereas change <0% is considered to be a decrease or a worse outcome. Subscales: The 3 subscales are: 1) knowledge of skin cancer, 2) risk factors, and 3) recognition of abnormal spots. The total number of correct answers are summed and divided by the total number of questions to calculate the total score.
Perceived importance, interest in, and confidence in looking for abnormal spots | 3 - 6 months
  Name of scale: Change in students' perceived importance, interest in, and confidence in looking for abnormal skin spots. What scale measures: Students selected from the following for perceived importance, interest in, and confidence in looking for abnormal skin spots: i)not at all; ii)slightly/a little bit; iii)somewhat; iv)definitely; or v) very/extremely important/interested in/confidence in (where i represents the lowest level and v represents the highest level). Self-reported post-tests were compared to pre-tests. If the amount of the self-reported importance, interest in or confidence was higher on the post-test compared to the pre-test, then it is considered an increase and a better outcome. Scale ranges: The change for perceived importance, interest in, and confidence in looking for abnormal skin spots were classified only as an increase (better outcome) or not (worse outcome).
Skin cancer risk behaviors | 3 - 6 months
  Name of scale: Change in indoor tanning, outdoor tanning, sunscreen and hat use. What scale measures: Students were asked to select from the following frequencies for tanning: 3-7 times per week, 1-2 times per week, 3-7 times in the last 2 months, 1-2 times in the last 2 months, none in the last 2 months. Students selected from the following for hat/sunscreen use: everyday, 1-6 times per week, 1-3 times per month, <1 time per month, or never. If the frequency of tanning was lower on the post-test compared to the pre-test, then it was classified as a decrease (which is a better outcome). If the frequency of sunscreen use/hat use was higher on the post-test compared to the pre-test, then it was classified as an increase (which is a better outcome). Scale range: The change for sunscreen/hat use was classified only as increasing (the better outcome) or not (the worse outcome); the change in tanning use was classified only as decreasing (the better outcome) or not (the worse outcome).
Communication with clients | 3 - 6 months
  Outcomes: Change in looking for abnormal skin spots, talking with clients about skin cancer prevention, and recommending a client see a doctor when an abnormal spot is seen. Students selected from the following proportion of clients in the last month they looked at for abnormal spots: none, <25%, 25-50%, 51-75%, or >75%; if the frequency for looking for abnormal spots reported on the post-test was greater than on the pre-test, then there was an increase (better outcome). Students also reported whether they discussed skin cancer prevention as either 'yes' or 'no', and whether or not they had ever recommended that a client see a doctor for an abnormal skin spot. Other outcomes were whether or not students reported on the post-test they looked for abnormal spots on >50% and >75% of their clients. Talking with clients about skin cancer prevention, and recommending a client see a doctor was increased (a better outcome) if they responded 'no' on the pre-test and 'yes' on the post-test.

CONTACTS AND LOCATIONS:
Overall Officials: Lori A Fischbach (co-Principal Investigator), PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No